CLINICAL TRIAL: NCT02038946
Title: A Single Arm, Open-Label Phase 2 Study of Nivolumab (BMS-936558) in Subjects With Relapsed or Refractory Follicular Lymphoma (FL)
Brief Title: Study of Nivolumab in Subjects With Relapsed or Refractory Follicular Lymphoma (FL) (CheckMate 140)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-140; 2013-003645-42 (EudraCT Number)
Record Dates: First submitted 2014-01-15; First posted 2014-01-17 (Estimated); Results first posted 2018-06-12 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1: Nivolumab (Experimental): Nivolumab 3 mg/kg injection by Intravenous for every 2 weeks until disease progression or discontinuation due to toxicity
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab
  Other Names: BMS-936558

SUMMARY:
The purpose of this study is to assess the clinical benefit of Nivolumab, as measured by independent radiologic review committee (IRRC)-assessed objective response rate (ORR) in subjects with FL lymphoma who have failed therapy with both CD20 antibody and an alkylating agent.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Grade 1, 2, or 3a FL without pathologic evidence of transformation
* Male and female, ages 18 and above, with relapsed or refractory FL lymphoma after > or =2 prior treatment lines; each of the 2 prior treatment lines must include at least CD20 antibody and/or an alkylating agent
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-1

Exclusion Criteria:

* Known central nervous system lymphoma
* History of interstitial lung disease
* Subjects with active, known or suspected autoimmune disease
* Prior allogeneic stem cell transplant
* Prior autologous stem cell transplant ≤12 weeks prior to first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2014-03-26 (Actual); Primary Completion 2017-05-17 (Actual); Study Completion 2020-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (44):
- United States (12):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Division Of Hematology & Oncology Ctr. For Health Sciences, Los Angeles, California
  - Winship Cancer Institute., Atlanta, Georgia
  - Beth Israel Deaconess Medical Center (BIDMC), Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Weill Cornell Medical College, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
- Australia (2):
  - Local Institution, Woodville, South Australia
  - Local Institution, Parkville, Victoria
- Belgium (3):
  - Local Institution, B-leuven
  - Local Institution, Brussels
  - Local Institution, Ghent
- Canada (2):
  - Jewish General Hospital, Montreal, Quebec
  - CISSS du Bas-Saint-Laurent Hopital Regional de Rimouski, Rimouski, Quebec
- France (4):
  - Local Institution, Créteil
  - Local Institution, Montpellier
  - Local Institution, Pierre-Bénite
  - Local Institution, Rennes
- Germany (5):
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum d. Saarlandes, Homburg
  - Universitaetsklinikum Des Saarlandes, Homburg
  - Local Institution, Regensburg
  - Universitaetsklinikum Ulm, Ulm
- Italy (5):
  - Local Institution, Bergamo
  - Local Institution, Bologna
  - Local Institution, Milan
  - Local Institution, Napoli
  - Local Institution, Roma
- Local Institution, Oslo, Norway
- Local Institution, Singapore, Singapore
- Spain (4):
  - Hospital Duran I Reynals, Hospitalet Llobregat- Barcelona
  - Local Institution, Madrid
  - Hospital Universitario La Paz, Madrid
  - Local Institution, Salamanca
- Sweden (2):
  - Local Institution, Gothenberg
  - Local Institution, Gothenburg
- United Kingdom (3):
  - Local Institution, Southampton, Hampshire
  - Local Institution, Withington, Manchester
  - Local Institution, Sutton, Surrey

REFERENCES:
- [Derived] Armand P, Janssens A, Gritti G, Radford J, Timmerman J, Pinto A, Mercadal Vilchez S, Johnson P, Cunningham D, Leonard JP, Rodig SJ, Martin-Regueira P, Sumbul A, Samakoglu S, Tang H, Ansell SM. Efficacy and safety results from CheckMate 140, a phase 2 study of nivolumab for relapsed/refractory follicular lymphoma. Blood. 2021 Feb 4;137(5):637-645. doi: 10.1182/blood.2019004753. PMID 32870269
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 116 participants were enrolled; 92 received study treatment. Participants were enrolled but not treated because they no longer met study criteria (n=20), withdrew consent (n=1), or for other reasons (n=3).
Groups:
- Arm 1: Nivolumab: Nivolumab 3mg/kg intravenously every 2 weeks until disease progression or discontinuation due to toxicity
Period: Overall Study
Arm/Group | Arm 1: Nivolumab
Started | 92
Completed (Completed = Participants continuing in the Follow-up period) | 80
Not Completed | 12
Not completed — Death | 5
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 2
Not completed — Other reasons | 2

BASELINE CHARACTERISTICS:
Population: All treated participants
Arm/Group | Arm 1: Nivolumab
Number analyzed (Participants) | 92
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: All treated participants
  years | 65.2 (10.50)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All treated participants
  Participants
    Female | 44
    Male | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: All treated participants
  Participants
    Hispanic or Latino | 5
    Not Hispanic or Latino | 49
    Unknown or Not Reported | 38
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: All treated participants
  Participants
    American Indian or Alaska Native | 0
    Asian | 3
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 1
    White | 87
    More than one race | 0
    Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) as Determined by IRRC
Description: ORR is determined by an independent radiologic review committee (IRRC) according to the revised International Working Group Criteria for non-Hodgkin Lymphoma. ORR is defined as the number of participants with a best overall response (BOR) of complete response (CR) or partial response (PR) and expressed as a percentage of all treated participants.
  CR=Disappearance of all clinical/radiographic evidence of disease, regression of lymph nodes to normal size, absence of spleen, liver, and bone marrow involvement.
  PR=Regression of measurable disease and no new sites; no increase in size of liver or spleen. >=50% decrease in SPD of up to 6 largest dominant masses (index lesions); no increase in size of other nodes (non-index lesions)
Time Frame: From Week 9 until documented disease progression or study discontinuation (assessed up to June 2017, approximately 38 months)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: Nivolumab
Number analyzed (Participants) | 92
Percentage of participants | 4.3 [1.2 to 10.8]

2. Secondary Outcome: Duration of Response (DOR) Based on IRRC Assessments
Description: DOR is defined as the time from first remission (CR or PR) to the date of initial objectively documented progression as determined using the revised International Working Group Criteria for non-Hodgkin Lymphoma, or death due to any cause, whichever occurs first.
  CR definition includes the complete disappearance of all evidence of disease, the definition of PR includes at least a 50% decrease in sum of the product of the diameters (SPD) of up to six of the largest dominant nodes or nodal masses, and PD is defined as any new lesion or increase by >50% of previously involved sites from nadir, as described in the IWG response criteria
Time Frame: as for outcome 1
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1: Nivolumab
Number analyzed (Participants) | 92
months | 10.94 [8.31 to 13.57]

3. Secondary Outcome: Complete Remission Rate (CRR) Based on IRRC Assessment
Description: CRR is defined as the number of subjects with a BOR of CR according to the revised International Working Group Criteria for non-Hodgkin Lymphoma, divided by the number of treated participants and expressed as a percentage.
  CR=Disappearance of all clinical/radiographic evidence of disease, regression of lymph nodes to normal size, absence of spleen, liver, and bone marrow involvement.
Time Frame: as for outcome 1
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: Nivolumab
Number analyzed (Participants) | 92
Percentage of participants | 1.1 [0.0 to 5.9]

4. Secondary Outcome: Partial Remission (PR) Rate Based on IRRC Assessment
Description: PR rate is defined as the number of participants with a best overall response (BOR) of PR according to the 2007 International Working Group (IWG) criteria, based on IRRC assessment, divided by the number of treated participants and expressed as a percentage.
  PR=Regression of measurable disease and no new sites; no increase in size of liver or spleen. >=50% decrease in SPD of up to 6 largest dominant masses (index lesions); no increase in size of other nodes (non-index lesions)
Time Frame: as for outcome 1
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: Nivolumab
Number analyzed (Participants) | 92
Percentage of participants | 3.3 [0.7 to 9.2]

5. Secondary Outcome: Progression Free Survival (PFS) Based on IRRC Assessment
Description: PFS was summarized descriptively using the Kaplan-Meier (KM) product-limit method. Median values of PFS, along with the two-sided 95% CIs were calculated using a method based on log-log transformation.
Time Frame: as for outcome 1
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1: Nivolumab
Number analyzed (Participants) | 92
months | 2.20 [1.91 to 3.58]

6. Secondary Outcome: Overall Response Rate (ORR) Based on Investigator Assessments
Description: ORR is determined by investigator assessments according to the revised International Working Group Criteria for non-Hodgkin Lymphoma. ORR is defined as the number of subjects with a best overall response (BOR) of complete response (CR) or partial response (PR) and is expressed as a percentage of all treated participants.
  CR=Disappearance of all clinical/radiographic evidence of disease, regression of lymph nodes to normal size, absence of spleen, liver, and bone marrow involvement.
  PR=Regression of measurable disease and no new sites; no increase in size of liver or spleen. >=50% decrease in SPD of up to 6 largest dominant masses (index lesions); no increase in size of other nodes (non-index lesions)
Time Frame: as for outcome 1
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: Nivolumab
Number analyzed (Participants) | 92
Percentage of participants | 10.9 [5.3 to 19.1]

ADVERSE EVENTS:
Time Frame: AEs collected were reported between first dose and 100 days after last dose of study therapy (up to approximately 6 years 9 months)
Groups:
- Nivolumab 3 mg/kg: Nivolumab 3mg/kg intravenously every 2 weeks until disease progression or discontinuation due to toxicity
Arm/Group | Nivolumab 3 mg/kg
All-Cause Mortality (participants affected / at risk) | 36/92
Serious Adverse Events (participants affected / at risk) | 46/92
Other Adverse Events (participants affected / at risk) | 89/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab 3 mg/kg (N=92)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1
Cytopenia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Pancytopenia (Blood and lymphatic system disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiac failure acute (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Ascites (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Fatigue (General disorders) | 1
General physical health deterioration (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Pyrexia (General disorders) | 6
Anaphylactic shock (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Appendicitis (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 2
Erysipelas (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 2
Lower respiratory tract infection (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 2
Pulmonary sepsis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 2
Staphylococcal sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Influenza B virus test positive (Investigations) | 1
Transaminases increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Sciatica (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Immune-mediated pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab 3 mg/kg (N=92)
Anaemia (Blood and lymphatic system disorders) | 15
Neutropenia (Blood and lymphatic system disorders) | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 8
Abdominal pain (Gastrointestinal disorders) | 15
Constipation (Gastrointestinal disorders) | 14
Diarrhoea (Gastrointestinal disorders) | 22
Dysphagia (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 23
Vomiting (Gastrointestinal disorders) | 12
Asthenia (General disorders) | 9
Fatigue (General disorders) | 23
Oedema peripheral (General disorders) | 10
Pyrexia (General disorders) | 25
Nasopharyngitis (Infections and infestations) | 8
Pneumonia (Infections and infestations) | 6
Upper respiratory tract infection (Infections and infestations) | 11
Urinary tract infection (Infections and infestations) | 9
Decreased appetite (Metabolism and nutrition disorders) | 14
Hypokalaemia (Metabolism and nutrition disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 11
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Dizziness (Nervous system disorders) | 7
Headache (Nervous system disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 25
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 11
Rash (Skin and subcutaneous tissue disorders) | 8
Skin lesion (Skin and subcutaneous tissue disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2016-07-21): https://cdn.clinicaltrials.gov/large-docs/46/NCT02038946/Prot_002.pdf
  • Statistical Analysis Plan (2017-06-27): https://cdn.clinicaltrials.gov/large-docs/46/NCT02038946/SAP_001.pdf